CLINICAL TRIAL: NCT05278390
Title: Automated Quantification of Radiologic Pulmonary Alteration During Acute Respiratory Failure: Application to the COVID-19 Pandemic : Prospective Multicenter Cohort Study
Brief Title: Automated Quantification of Radiologic Pulmonary Alteration During Acute Respiratory Failure: Application to the COVID-19 Pandemic
Acronym: QUANTICO-PRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: REGION GRAND EST (Unknown); E-MEDIA (Unknown); VISIBLE PATIENT (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8138
Record Dates: First submitted 2022-03-11; First posted 2022-03-14 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: SARS-CoV-2 Infections; Respiratory Failure With Hypoxia
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thoracic CT Scan (Experimental)
  Interventions: Radiation: Thoracic CT scan

INTERVENTIONS:
Radiation: Thoracic CT scan — Automated quantitative analysis of altered pulmonary volume

SUMMARY:
Automated quantification of the pulmonary volume impaired during acute respiratory failure could be helpful to assess patient severity during COVID-19 infection or perioperative medicine, for example.

This study aims at assessing the correlation between the amount of radiologic pulmonary alteration and the clinical severity in two clinical situation :

1. SARS-CoV-2 infections
2. Postoperative hypoxemic acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Subject admitted to a care unit of the University Hospitals of Strasbourg or the University Hospital of Nancy and presenting a suspicion of SARS-CoV-2 infection or postoperative hypoxemic respiratory failure
* Able to understand the objectives and risks of the research and to give dated and signed informed consent.

Subjects may also be included in emergency or immediate life-threatening situations.

* Subject with insurance covering

Exclusion Criteria:

* Pregnant woman (pregnancy confirmed by a urine or blood test)
* Subject usually on home oxygen therapy
* Subject under court protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between altered pulmonary volume and ordinal severity scale | 2 days after CT scan (Day 2)
  This criterion will be expressed as a score between 1 (least severe) and 7 (most severe).

SECONDARY OUTCOMES:
Correlation between altered pulmonary volume and ordinal severity scale | 7 days after CT scan (Day 7)
  This criterion will be expressed as a score between 1 (least severe) and 7 (most severe).
Mortality | 90 days following CT scan (Day 90)
Rate of admission to intensive care unit | 28 days following CT scan (Day 28)
Initial length of hospitalization stay (in days) | 90 days following CT scan (Day 90)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service d'anesthésie réanimation-CHU de Nancy, Nancy
  - Service d'Anesthésie-Réanimation - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No